CLINICAL TRIAL: NCT06244667
Title: Comparison of Different Local Anesthetics in Cervical Facet Medial Branch Blockade
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ankara University (Other)
Responsible Party: Principal Investigator, Hanzade Aybuke Unal, Director, Ankara University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2023/468
Record Dates: First submitted 2024-01-20; First posted 2024-02-06 (Actual); Last update posted 2024-02-06 (Actual); Status verified 2024-01

CONDITIONS: Pain, Neck
Keywords: pain; nerve block
MeSH Terms: conditions — Neck Pain; Pain | interventions — Prilocaine; Lidocaine

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- cervical faset median block with lidocaine (Active Comparator): cervical faset median block with lidocaine
  Interventions: Procedure: facet median block with lidocaine
- cervical faset median block with prilocaine (Active Comparator): cervical faset median block with prilocaine
  Interventions: Procedure: facet median block with prilocain

INTERVENTIONS:
Procedure: facet median block with prilocain — facet median block with prilocain
  Arms: cervical faset median block with prilocaine
Procedure: facet median block with lidocaine — facet median block with lidocaine
  Arms: cervical faset median block with lidocaine

SUMMARY:
Neck pain is a common disease in society. In studies, the annual and lifetime prevalence was found to be 37.2% and 48.5%, respectively (1). Neck pain may be axial or radicular. Causes of axial neck pain include cervical strain, discogenic pain, cervical facet pain, spondylosis, whiplash, and myofascial pain. (2) Cervical facet degeneration is a common cause of axial neck pain (3). Pain originating from the cervical facet joint is localized to the midline of the neck and increases with neck extension. (2) Diagnosis is made by physical examination and radiological imaging. The distribution patterns of pain originating from the cervical facet joint vary depending on the level of the joint involved

DETAILED DESCRIPTION:
Neck pain is a common disease in society. Causes of axial neck pain include cervical strain, discogenic pain, cervical facet pain, spondylosis, whiplash, and myofascial pain. Cervical facet degeneration is a common cause of axial neck pain. Pain originating from the cervical facet joint is localized to the midline of the neck and increases with neck extension. Diagnosis is made by physical examination and radiological imaging. The distribution patterns of pain originating from the cervical facet joint vary depending on the level of the joint involved.

Conservative treatment methods for facet joint pain are medical treatment and various physical therapy modalities. Interventional pain treatments are on the agenda for patients who cannot achieve effective pain palliation with conservative treatment. Since facet joints are innervated by the dorsal ramus, medial branch of the spinal nerves, medial branch blockade is applied in the treatment of facet-related pain. In cervical facet medial branch blockade, a mixture of local anesthetic and steroid is injected. Studies have found that adding steroids to local anesthetics increases injection effectiveness. Although there is no consensus on the type of steroid to be used, it is safer to use dexamethasone, a particle-free steroid, considering the dense vascular structure of the cervical region. However, the types of local anesthetic used in cervical facet medial branch blockade vary between studies. The type of local anesthetic used in cervical facet medial branch blockade in our clinic varies. There is only one study in the literature comparing local anesthetic types. Researchers compared the effectiveness of lidocaine and bupivacaine in cervical facet medial branch blockade without adding steroids. Researchers stated that lidocaine has a faster effect and longer duration of effect. Since there is no consensus on the type of local anesthetic, prilocaine or lidocaine is preferred in practice. This study aims to compare the effectiveness of lidocaine and prilocaine added to dexamethasone in cervical facet medial branch blockade, one of the routine treatment methods in our clinic.

Within the scope of the study, patients deemed suitable for cervical facet medial branch injection will be randomly numbered for prilocaine or lidocaine injection through the computer program. 57 patients will receive lidocaine + steroid injection, 57 patients will receive prilocaine + steroid injection. Cervical facet medial branch injections will be administered. The evaluations of the patients before and after the procedure will be recorded by the researcher who is blind to the procedure performed. Demographic information of the patients, including age, gender, comorbidities, pain duration, and facet injection level, will be recorded before the procedure. Before the procedure, pain intensity will be evaluated using the NRS 11 scale, and functionality will be evaluated using the Neck Disability Index (NDI). The amount of medication used by the patients (non-steroidal anti-inflammatory analgesics, opioids, muscle relaxants) will also be noted.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 20-79
* A history of axial cervical pain without radicular symptoms for at least 3 months
* NRS score of 4 and above
* Not having had a cervical interventional procedure in the last year
* Patients who cannot achieve adequate pain palliation with pharmacological and physical treatment modalities

Exclusion Criteria:

* Patients experiencing cervical radicular pain due to disc herniation or foraminal stenosis and neck pain due to cervical canal stenosis
* Patients with previous cervical surgery
* Patients with psychiatric illnesses that are unstable/uncontrolled with medical treatment
* Pregnant patients
* Bleeding diathesis
* Patients who received epidural steroid injection within the last year
* Patients with known allergies to the substances administered during the procedure (local anesthetic, steroid, contrast material)
* Patients with cervical spondylosis, radiculopathy, myelopathy, spondylolisthesis, compression fracture, previous discitis, sequestered disc, overt disc herniation

Ages: 20 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 114 (Actual)
Dates: Start 2023-10-01 (Actual); Primary Completion 2024-01-01 (Actual); Study Completion 2024-01-01 (Actual)

PRIMARY OUTCOMES:
change of pain intensity | 1 month
  Change from baseline in pain scores on the Numeric Rating Scale at 1 month in both groups
change of participants functionality | 1 month
  Change of participants functionality (Neck Disability Score) at 1 month in both groups
participants satisfaction | 1 month
  Participants satistification degree (satisfied", "uncertain" or "dissatisfied") at 1 month in both groups

SECONDARY OUTCOMES:
drug use in groups | 1 month
  the effect of lidocaine and prilocaine injection applied in addition to dexamethasone in cervical facet medial blockade on drug use.
difference of drug use between groups | 1 month
  the effect of lidocaine and prilocaine injection applied in addition to dexamethasone in cervical facet medial blockade on drug use.

CONTACTS AND LOCATIONS:
Overall Officials: Gungor E Özgencil, Prof, Study Director — Ankara University
Locations (1):
- Ankara University, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Manchikanti L, Singh V, Falco FJ, Cash KM, Fellows B. Cervical medial branch blocks for chronic cervical facet joint pain: a randomized, double-blind, controlled trial with one-year follow-up. Spine (Phila Pa 1976). 2008 Aug 1;33(17):1813-20. doi: 10.1097/BRS.0b013e31817b8f88. PMID 18670333
- [Background] Manchikanti L, Sanapati MR, Pampati V, Soin A, Atluri S, Kaye AD, Subramanian J, Hirsch JA. Update of Utilization Patterns of Facet Joint Interventions in Managing Spinal Pain from 2000 to 2018 in the US Fee-for-Service Medicare Population. Pain Physician. 2020 Mar;23(2):E133-E149. PMID 32214289